CLINICAL TRIAL: NCT02776930
Title: Development of Predictive Models for Lower Extremity, Lumbar, and Thoracic Injury After Discharge From Physical Rehabilitation
Brief Title: Predictive Models for Spine and Lower Extremity Injury After Discharge From Rehab
Acronym: MP3-RD
Status: Completed | Type: Observational
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Collaborators: Womack Army Medical Center (U.S. Federal Agency); William Beaumont Army Medical Center (U.S. Federal Agency); Madigan Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dan Rhon, Director of Physical Therapy, Center for the Intrepid, Brooke Army Medical Center
Other Study IDs: 215032
Record Dates: First submitted 2016-05-17; First posted 2016-05-18 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Musculoskeletal Injury; Spinal Injuries; Leg Injuries
Keywords: Injury Prediction; Return to Work; Injury Prevention
MeSH Terms: conditions — Spinal Injuries; Leg Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Return to Duty after Rehab from Injury: Patients deemed healthy enough to return to full duty without any restrictions after completing a course of rehabilitation for a lumbar/thoracic spine or lower extremity injury.

SUMMARY:
The purpose of this study is to develop algorithms that will help predict future injury and/or re-injury after being returned to duty from a musculoskeletal injury. After completion of an episode of care with a physical therapist, the subjects will undergo a battery of physical performance tests and fill out associated surveys. The subjects will then be followed for a year to identify the occurrence/re-occurence of any injuries. Based on the performance on the physical evaluation tests, algorithms will be derived using regression analysis to predict injury.

Subjects will be recruited from the pool of patients that have recently completed physical rehabilitation in physical therapy clinics for their lower extremity or lumbar/thoracic spine injury.

DETAILED DESCRIPTION:
Subjects will be recruited across 4 medical centers after having completed a regimen of physical therapy for a spine or lower extremity injury. Upon discharge back to full duty, they will be given the opportunity to enroll in the study and undergo a battery of physical performance tests and associated surveys. The subjects will then be followed for a year to identify the occurrence of any injuries. Prediction algorithms will be derived using regression analysis to predict injury based on performance on the physical evaluation tests.

The overall hypothesis is that Service Member performance on a battery of physical performance tests performed upon discharge from care and return to duty, will be able to predict 1) the risk of sustaining any injury as well as 2) reoccurrence of the same injury that they were seeking care for during the year following discharge from rehabilitation. The current assumption is that when a Service Member is discharged from medical care, it has been done based on the expectation that it is appropriate and safe for them to return to function in their operational environment. Because history of prior injury is a well-established risk factor, every single Service Member that is returned to duty after medical care for a musculoskeletal (MSK) injury is already at a higher risk for future injury than his or her non-injured counterpart. The investigators hypothesize that decreased performance on the proposed testing protocol will be related to increase in the risk of 1 year-injury and recurrence of injury. Successfully identifying those at increased risk of recurrence provides the ability for secondary and tertiary prevention programs to optimize return to duty rates. Injury will be defined as any new musculoskeletal injury or the re-occurrence of the same injury during the 1-year surveillance period.

The battery of physical performance tests will include: Selective Functional Movement Assessment (SFMA), Functional Movement Screen (FMS), Upper Quarter Y-balance Test (YBT-UQ), Lower Quarter Y-balance Test (YBT-LQ), Closed Kinetic Chain Dorsiflexion (CKC DF), a Single Hop Test, Triple Hop Test, Triple Crossover Hop Test, Carry Test, and a un-weighted and weighted 300 yard Shuttle Run Test.

Each subject will then also be contacted monthly via a SMS (Short Message Service, e.g. text message) survey for the following year to identify information about additional injury or profile that they may have sustained during the prior period of time. Information about injury will also be calculated from patient chart reviews and Department of Defense healthcare utilization database (claims data). This will provide a robust method in which to capture data injury data regardless of subject availability for follow-up.

Subjects will be dichotomized as injured or non-injured based on the injury surveillance data. Key demographic, physical performance (FMS, YBT, SFMA, Hop Test, Carry test, & Shuttle Run), and self-report measures will be examined for group differences. Potential predictor variables will be entered into a backward stepwise logistic regression model to determine the most accurate set of variables predictive of musculoskeletal injury status.

Risk stratification (low, moderate, or high) will be based on likelihood ratios (LR) associated with the clinical prediction rule for injury outlined above. A positive LR > 10 will place the individual as high risk, a LR between 2 and 10 would place the individual as moderate risk. Those with a positive LR less than 2 will be listed as low risk.

ELIGIBILITY:
Inclusion Criteria:

1. Active duty service member eligible for Tricare benefits
2. Lower extremity or lumbar/thoracic spine injury is the patient's primary complaint.
3. Determined fit for duty (cleared to return to work) after completing a course of physical therapy for a lower extremity or lumbar/thoracic spine musculoskeletal injury

Exclusion Criteria:

1. Individuals planing on leaving the military within the next 10 months.
2. Trauma or polytrauma that results in amputation of any limbs or appendages.
3. Pregnancy, or recently pregnant within the last 6 months - subjects that become pregnant during the course of the study will be withdrawn based on the different injury risk factors that are associated with pregnancy.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Active duty service members that have completed a course of physical therapy for a spine or lower extremity injury, and then discharged to return to full duty.
Sampling Method: Non-Probability Sample
Enrollment: 480 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-09-19 (Actual); Study Completion 2019-11-19 (Actual)

PRIMARY OUTCOMES:
Injury Occurrence | 1 year
  Monthly SMS survey capturing new musculoskeletal injury since the prior survey

SECONDARY OUTCOMES:
Injury-Related Healthcare Utilization | 1 year
  Healthcare utilization for musculoskeletal injury taken from the Tricare claims database (MHS Data Repository)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Rhon, DSc, Principal Investigator — Brooke Army Medical Center
Locations (4):
- United States (4):
  - Womack Army Medical Center, Fort Bragg, North Carolina
  - William Beaumont Army Medical Center, Fort Bliss, Texas
  - Brooke Army Medical Center, San Antonio, Texas
  - Madigan Army Medical Center, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing must be requested and approved through the Defense Health Agency via a Data Sharing Agreement Application

REFERENCES:
- [Background] Lincoln AE, Smith GS, Amoroso PJ, Bell NS. The natural history and risk factors of musculoskeletal conditions resulting in disability among US Army personnel. Work. 2002;18(2):99-113. PMID 12441574
- [Background] Ernat J, Knox J, Orchowski J, Owens B. Incidence and risk factors for acute low back pain in active duty infantry. Mil Med. 2012 Nov;177(11):1348-51. doi: 10.7205/milmed-d-12-00183. PMID 23198512
- [Background] Knapik JJ, Graham B, Cobbs J, Thompson D, Steelman R, Jones BH. A prospective investigation of injury incidence and injury risk factors among Army recruits in military police training. BMC Musculoskelet Disord. 2013 Jan 17;14:32. doi: 10.1186/1471-2474-14-32. PMID 23327563
- [Background] Jones BH, Thacker SB, Gilchrist J, Kimsey CD Jr, Sosin DM. Prevention of lower extremity stress fractures in athletes and soldiers: a systematic review. Epidemiol Rev. 2002;24(2):228-47. doi: 10.1093/epirev/mxf011. No abstract available. PMID 12762095
- [Background] Wilkinson DM, Blacker SD, Richmond VL, Horner FE, Rayson MP, Spiess A, Knapik JJ. Injuries and injury risk factors among British army infantry soldiers during predeployment training. Inj Prev. 2011 Dec;17(6):381-7. doi: 10.1136/ip.2010.028233. Epub 2011 Apr 19. PMID 21507884
- [Background] Lehr ME, Plisky PJ, Butler RJ, Fink ML, Kiesel KB, Underwood FB. Field-expedient screening and injury risk algorithm categories as predictors of noncontact lower extremity injury. Scand J Med Sci Sports. 2013 Aug;23(4):e225-32. doi: 10.1111/sms.12062. Epub 2013 Mar 20. PMID 23517071
- [Background] Butler RJ, Contreras M, Burton LC, Plisky PJ, Goode A, Kiesel K. Modifiable risk factors predict injuries in firefighters during training academies. Work. 2013 Jan 1;46(1):11-7. doi: 10.3233/WOR-121545. PMID 23324700
- [Background] Peate WF, Bates G, Lunda K, Francis S, Bellamy K. Core strength: a new model for injury prediction and prevention. J Occup Med Toxicol. 2007 Apr 11;2:3. doi: 10.1186/1745-6673-2-3. PMID 17428333
- [Background] Larsson H, Broman L, Harms-Ringdahl K. Individual risk factors associated with premature discharge from military service. Mil Med. 2009 Jan;174(1):9-20. doi: 10.7205/milmed-d-03-7407. PMID 19216293
- [Background] Bahr R. Why screening tests to predict injury do not work-and probably never will...: a critical review. Br J Sports Med. 2016 Jul;50(13):776-80. doi: 10.1136/bjsports-2016-096256. Epub 2016 Apr 19. PMID 27095747
- [Result] Jones BH, Perrotta DM, Canham-Chervak ML, Nee MA, Brundage JF. Injuries in the military: a review and commentary focused on prevention. Am J Prev Med. 2000 Apr;18(3 Suppl):71-84. doi: 10.1016/s0749-3797(99)00169-5. PMID 10736543
- [Result] Knapik JJ, Bullock SH, Canada S, Toney E, Wells JD, Hoedebecke E, Jones BH. Influence of an injury reduction program on injury and fitness outcomes among soldiers. Inj Prev. 2004 Feb;10(1):37-42. doi: 10.1136/ip.2003.002808. PMID 14760025
- [Result] Parkkari J, Kujala UM, Kannus P. Is it possible to prevent sports injuries? Review of controlled clinical trials and recommendations for future work. Sports Med. 2001;31(14):985-95. doi: 10.2165/00007256-200131140-00003. PMID 11735682
- [Result] de la Motte SJ, Lisman P, Sabatino M, Beutler AI, O'Connor FG, Deuster PA. The Relationship Between Functional Movement, Balance Deficits, and Previous Injury History in Deploying Marine Warfighters. J Strength Cond Res. 2016 Jun;30(6):1619-25. doi: 10.1519/JSC.0000000000000850. PMID 26964060
- [Result] Kodesh E, Shargal E, Kislev-Cohen R, Funk S, Dorfman L, Samuelly G, Hoffman JR, Sharvit N. Examination of the Effectiveness of Predictors for Musculoskeletal Injuries in Female Soldiers. J Sports Sci Med. 2015 Aug 11;14(3):515-21. eCollection 2015 Sep. PMID 26336337
- [Result] Bonazza NA, Smuin D, Onks CA, Silvis ML, Dhawan A. Reliability, Validity, and Injury Predictive Value of the Functional Movement Screen: A Systematic Review and Meta-analysis. Am J Sports Med. 2017 Mar;45(3):725-732. doi: 10.1177/0363546516641937. Epub 2016 Jul 21. PMID 27159297
- [Derived] Rhon DI, Plisky PJ, Kiesel K, Greenlee TA, Bullock GS, Shaffer SW, Goffar SL, Teyhen DS. Predicting Subsequent Injury after Being Cleared to Return to Work from Initial Lumbar or Lower Extremity Injury. Med Sci Sports Exerc. 2023 Dec 1;55(12):2115-2122. doi: 10.1249/MSS.0000000000003257. Epub 2023 Jul 27. PMID 37486770
- [Derived] Rhon DI, Teyhen DS, Shaffer SW, Goffar SL, Kiesel K, Plisky PP. Developing predictive models for return to work using the Military Power, Performance and Prevention (MP3) musculoskeletal injury risk algorithm: a study protocol for an injury risk assessment programme. Inj Prev. 2018 Feb;24(1):81-88. doi: 10.1136/injuryprev-2016-042234. Epub 2016 Nov 24. PMID 27884941